CLINICAL TRIAL: NCT05306158
Title: Approach Bias Retraining for Nicotine Addiction Among Dual Combustible and Electronic Cigarette Users
Brief Title: Dual Use Approach Bias Training for Nicotine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Lorra Garey, Assistant Research Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR-19-309
Record Dates: First submitted 2022-02-16; First posted 2022-03-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Smoking; Electronic Cigarette Use; Substance Use
MeSH Terms: conditions — Tobacco Smoking; Vaping; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: There are three arms, one intervention (CC+ECIG Condition), one active comparator (CC Condition), and one Sham (control) arm which are randomly assigned at the same time (baseline) and are implemented in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CC+ECIG Condition (Experimental): Combustible Cigarette (CC) and Electronic Cigarette (ECIG) users will be trained to avoid CC and ECIG-related images and approach positive images.
  Interventions: Other: CC+ECIG Condition
- CC Only Condition (Active Comparator): Participants in this arm will be trained to avoid only combustible cigarette images, not electronic cigarettes images.
  Interventions: Other: CC Condition
- Sham Condition (Sham Comparator): Participants will pull and push all pictures of CC and ECIG images equally with no preference towards one or the other.
  Interventions: Other: Sham Condition

INTERVENTIONS:
Other: CC+ECIG Condition — Participants will push CC- and ECIG-related pictures.
  Arms: CC+ECIG Condition
Other: CC Condition — Participants will push CC-related images and push and pull ECIG-related pictures equally often.
  Arms: CC Only Condition
Other: Sham Condition — Participants will pull and push CC- and ECIG-related pictures equally often.
  Other Names: Control
  Arms: Sham Condition

SUMMARY:
The present project will evaluate the initial efficacy of approach bias retraining among dual combustible cigarette (CC) and electronic cigarette (ECIG) users. The study employs a randomized controlled design to follow 90 experienced dual CC/ECIG users motivated to quit nicotine as they engage in a self-guided quit attempt following approach bias retraining.

DETAILED DESCRIPTION:
The study employs a randomized controlled design to follow 90 experienced dual CC/ECIG users motivated to quit nicotine as they engage in a self-guided quit attempt following approach bias retraining. Participants will be randomized to one of three approach bias retraining conditions: (1) CC+ECIG; (2) CC only; or (3) sham (control). Participants will complete a phone pre-screener, baseline (week 1 of study participation), 4 approach bias retraining sessions in laboratory (with quit day scheduled for the 4th session; weeks 2-5 of study participation), and follow-up assessments at 4- and 6-weeks post-intervention (i.e., weeks 9 and 11 of study participation, respectfully). Participants also will complete ecological momentary assessments (EMA) of CC smoking, ECIG use, and CC and ECIG urges/cravings for 14 days post-intervention (i.e., weeks 5-7 of study participation) on Internet capable smartphones. The only time data will be collected is when participants complete EMA assessments or follow up surveys using the REDCap app on the smartphone.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* At least 15 days of CC use for the previous month
* ECIG use with nicotine at least 15 days for the previous month
* Motivation to quit nicotine (BOTH CC and ECIG; ≥ 5 on a 0-10 scale)
* Ability to speak and read English fluently
* Not have decreased number of cigarettes by more than half in the past month
* Own an android smartphone (for EMA).

Exclusion Criteria:

* Current psychotherapy or pharmacotherapy for mental illness or addiction
* Current use of nicotine replacement therapy, Zyban, or Chantix
* Limited mental capacity or inability to provide informed consent
* Insufficient command of the English language (>6th grade English literacy level required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Biochemically-Verified Point Prevalence Abstinence | Week 9 of participation
  Biochemically-verified (urine and/or expired carbon monoxide reading) and self-reported 7-day abstinence prior to follow up (CC and/or ECIG)
Prolonged Abstinence | Week 9 of participation
  Smoking on fewer than 7 consecutive days or smoking fewer than once each week over 2 consecutive weeks (CC and/or ECIG)
Lapse | Week 9 of participation
  Time to first use (CC and/or ECIG)
Nicotine Relapse | Week 9 of participation
  7th day on which CC or ECIG occurs

SECONDARY OUTCOMES:
Questionnaire of Smoking Urges-Brief (QSU-Brief) | Week 1-7, 9, and 11 of participation
  The Brief Questionnaire of Smoking Urges (QSU-Brief) consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now).
Questionnaire of Vaping Craving | Week 1-7, 9, and 11 of participation
  The Questionnaire of Vaping Craving is a modified measure of the QSU and consists of 10 statements about the respondent's feelings and thoughts about his or her desire to vape as he or she is completing the questionnaire (i.e., right now).
Approach Bias | Weeks 2-5 of participation
  The approach-avoidance task (AAT) is a 15-minute computerized task instructs participants to use a joystick to either pull toward themselves or push away from themselves images presented on the screen that vary in content (i.e., substance-related, neutral, positive) and format (e.g., right- or left-tilted).
Biochemically-Verified Point Prevalence Abstinence | Week 11 of participation
  Biochemically-verified (urine and/or expired carbon monoxide reading) and self-reported 7-day abstinence prior to follow up (CC and/or ECIG)
Prolonged Abstinence | Week 11 of participation
  Smoking on fewer than 7 consecutive days or smoking fewer than once each week over 2 consecutive weeks (CC and/or ECIG)
Lapse | Week 11 of participation
  Time to first use (CC and/or ECIG)
Nicotine Relapse | Week 11 of participation
  7th day on which CC or ECIG occurs

CONTACTS AND LOCATIONS:
Overall Officials: Lorra Garey, Ph.D, Principal Investigator — Assistant Research Professor
Locations (1):
- RESTORE Laboratory, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide de-identified data from this project to interested individuals one year following achievement of the aims of the project (i.e., publication of the main outcome paper). These data will be provided in digital format (i.e., disk) with clear labels for all variables. Data will be released directly by the investigators providing evidence of their institution's IRB approval for planned analyses of the data. Our team will be available to address queries.
Supporting Information: Study Protocol, SAP
Time Frame: One year after completion upon request.
Access Criteria: Upon specific IRB approval and request from researchers.

REFERENCES:
- [Derived] Clausen B, Rinck M, Nizio P, Matoska CT, Zappi C, Smits JAJ, Gallagher MW, Zvolensky MJ, Garey L. Study protocol for approach bias retraining for nicotine addiction among dual combustible and electronic cigarette users. Contemp Clin Trials. 2023 May;128:107145. doi: 10.1016/j.cct.2023.107145. Epub 2023 Mar 9. PMID 36905980